CLINICAL TRIAL: NCT03012061
Title: A Phase IIb, 24 Week, Randomized, Double-blind, 3 Arm Parallel Group Study, Comparing the Efficacy, Safety and Tolerability of Two Doses of Umeclidinium Bromide Administered Once-daily Via a Dry Powder Inhaler, Versus Placebo, in Participants With Asthma
Brief Title: Phase IIb Study of Umeclidinium (UMEC) Bromide Versus Placebo in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205832; 2016-002843-40 (EudraCT Number)
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: Respiratory; Efficacy; Umeclidinium bromide; Parallel; Asthma; Dry powder inhaler
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects will be administered placebo once daily via the ELLIPTA® dry powder inhaler (DPI) for 24 weeks. Subjects will also receive FF 100 mcg once daily, in the morning for 24 weeks. ELLIPTA is a registered trademark of the GSK group of companies.
  Interventions: Drug: Placebo; Drug: Fluticasone Furoate; Drug: Albuterol/salbutamol
- UMEC 62.5 mcg (Experimental): Subjects will be administered UMEC 62.5 mcg once daily via the ELLIPTA dry powder inhaler (DPI) for 24 weeks. Subjects will also receive FF 100 mcg once daily, in the morning for 24 weeks.
  Interventions: Drug: UMEC; Drug: Fluticasone Furoate; Drug: Albuterol/salbutamol
- UMEC 31.25 mcg (Experimental): Subjects will be administered UMEC 31.25 mcg once daily via the ELLIPTA dry powder inhaler (DPI) for 24 weeks. Subjects will also receive FF 100 mcg once daily, in the morning for 24 weeks.
  Interventions: Drug: UMEC; Drug: Fluticasone Furoate; Drug: Albuterol/salbutamol

INTERVENTIONS:
Drug: Placebo — Placebo is a white powder to be administered using ELLIPTA DPI which hold two individual blister strips, both of which contains lactose monohydrate blended with magnesium stearate.
  Arms: Placebo
Drug: UMEC — UMEC is a white powder to be administered using ELLIPTA DPI which hold two individual blister strips, one of which contains GSK573719 blended with lactose blended with magnesium stearate and another one contains lactose monohydrate blended with magnesium stearate.
  Arms: UMEC 31.25 mcg; UMEC 62.5 mcg
Drug: Fluticasone Furoate — FF is a white powder to be administered using ELLIPTA DPI which hold two individual blister strips, one of which contains GW685698 blended with lactose monohydrate and another one contains lactose monohydrate with magnesium stearate.
Drug: Albuterol/salbutamol — Albuterol/salbutamol is to be administered via metered-dose inhaler as a rescue drug on need basis throughout the study.

SUMMARY:
This study is conducted to evaluate the effects of UMEC 62.5 microgram (mcg) and UMEC 31.25 mcg on lung function versus placebo after 24 weeks of treatment. This study will provide important information regarding the efficacy and safety of UMEC when administered in a separate inhaler to subjects on a background of fluticasone furoate (FF). This is a Phase IIb, randomized, double-blind, placebo controlled study that will compare the efficacy, safety and tolerability of UMEC (62.5 mcg and 31.25 mcg) administered once-daily in subjects with asthma that is not well controlled. Eligible subjects will be requested to participate in the study for a maximum of approximately 31 weeks with 4 phases (pre screening, screening/run-in, randomization/treatment and safety follow-up). The total number of randomized subjects required is approximately 384, with 128 subjects randomized 1:1:1 to each of the 3 double-blind treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of signing the informed consent.
* Subjects with a diagnosis of asthma as defined by the National Institutes of Health at least 6 months prior to Visit 0.
* Asthma Control Questionnaire (ACQ)-6 total score of >0.75 at Visit 1.
* Subjects are eligible if they have required daily Inhaled Corticosteroids (ICS) therapy >=100 milligram per day (mg/day) fluticasone propionate (FP) or equivalent with or without Long-Acting Beta-2-Agonists (LABA) or Long-Acting Muscarinic Antagonist (LAMA) for at least 12 weeks prior to Visit 0 and there have been no changes in maintenance asthma medications during the 4 weeks immediately prior to Visit 0. Dosing regimen (once or twice daily to equal the total daily dose) should be restricted to the current local product labels.
* A best pre-bronchodilator morning FEV1 <=85% of the predicted normal value. Predicted values will be based upon the European Respiratory Society (ERS) Global Lung Function Initiative. A best post-bronchodilator FEV1/ forced vital capacity (FVC) >=0.7 at Visit 1.
* Airway reversibility is defined as >=12% and >=200 mL increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol at Visit 1. Note: If the subject does not meet the above reversibility criteria at Visit 1 then the reversibility assessment may be repeated once within 7 days of Visit 1 if either criteria are met: The >=9% increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol at Visit 1; Documented evidence of a reversibility assessment within 1 year prior to Visit 1 which demonstrated a post-bronchodilator increase in FEV1 of >=12% and >=200 milliliter (mL). Should the subject successfully demonstrate airway reversibility (defined as >=12% and >=200 mL increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol) at the second attempt then, provided that all other eligibility criteria assessed at Visit 1 are met, the subject may enter the 2-week run-in period.
* All subjects must be able to replace their current Short-Acting Beta-2-Agonists (SABA) inhaler with albuterol/salbutamol aerosol inhaler at Visit 1 as needed for the duration of the study. Subjects must be judged capable of withholding albuterol/salbutamol for at least 6 hours prior to study visits.
* Both male and female subjects are eligible to participate in the study. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 5 days after the last dose of study treatment.
* Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form and in this protocol. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.

Inclusion Criteria (for randomization)

* ACQ-6 total score of >0.75 at Visit 2.
* Spirometry: A best pre-bronchodilator morning FEV1 <=85% of the predicted normal value at Visit 2. Predicted values will be based upon the ERS Global Lung Function Initiative.
* Alanine aminotransferase (ALT) <=2 x upper limit of normal (ULN). Alkaline phosphatase <=1.5 x ULN. Bilirubin <=1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Compliance with completion of the Daily electronic diary (eDiary) reporting defined as completion of all questions/assessments on >=4 of the last 7 days during the run-in period.

Exclusion Criteria:

* Chest X-ray documented pneumonia in the 12 weeks prior to Visit 1.
* Any severe asthma exacerbation, defined as deterioration of asthma requiring the use of systemic corticosteroids (oral, parenteral or depot) within 12 weeks of Visit 1, or an inpatient hospitalization or emergency department visit due to asthma that required systemic corticosteroids within 12 weeks of Visit 1.
* Current evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, lung cancer, or other respiratory abnormalities other than asthma.
* Women who are pregnant or lactating or are planning to become pregnant during the study.
* Immune suppression (e.g., Human Immunodeficiency Virus [HIV], Lupus) or other risk factors for pneumonia (e.g., neurological disorders affecting control of the upper airway, such as Parkinson's disease, Myasthenia Gravis). Subjects at potentially high risk (e.g., very low Body Mass Index [BMI], severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator
* Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Chronic stable hepatitis B and C is acceptable if the subject otherwise meets entry criteria.
* Evidence of a clinically significant abnormality in the 12-lead ECG performed during screening or run-in. The Principal Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: Atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute (BPM); Sustained or nonsustained ventricular tachycardia (VT); Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 millisecond (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.
* Subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure.
* Subjects with a medical condition such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction should only be included if in the opinion of the Investigator the benefit outweighs the risk and that the condition would not contraindicate study participation.
* Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Subjects who are medically unable to withhold their albuterol/salbutamol for the 6-hour period required prior to spirometry testing at each study visit.
* Current smoker or a smoking history of >=10 pack years (e.g., 20 cigarettes/day for 10 years). A subject may not have used inhaled tobacco products within the past 12 months (i.e., cigarettes, e-cigarettes/vaping, cigars or pipe tobacco).
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years. This includes marijuana, which is considered an abused drug.
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate.
* Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.

Exclusion Criteria (for randomization)

* Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Evidence of a moderate asthma exacerbation leading to a change in therapy or severe exacerbation during screening or the run-in period, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Changes in asthma medication (excluding changes after Visit 0 or run-in medication and albuterol/salbutamol inhalation aerosol provided at Visit 1).
* Evidence of clinically significant abnormal laboratory tests during screening or run-in, which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (65):
- United States (18):
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Monroe, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Old Point Station, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Dallas, Texas
- Canada (10):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Corunna, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Poland (13):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zgierz
- Romania (10):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Sibiu
  - GSK Investigational Site, Timișoara
- Russia (14):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Odintsovo
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Volgodonsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20592

REFERENCES:
- [Background] Kerwin E, Pascoe S, Bailes Z, Nathan R, Bernstein D, Dahl R, von Maltzahn R, Robbins K, Fowler A, Lee L. A phase IIb, randomised, parallel-group study: the efficacy, safety and tolerability of once-daily umeclidinium in patients with asthma receiving inhaled corticosteroids. Respir Res. 2020 Jun 12;21(1):148. doi: 10.1186/s12931-020-01400-5. PMID 32532275
- [Derived] Oppenheimer J, Hanania NA, Chaudhuri R, Sagara H, Bailes Z, Fowler A, Peachey G, Pizzichini E, Slade D. Clinic vs Home Spirometry for Monitoring Lung Function in Patients With Asthma. Chest. 2023 Nov;164(5):1087-1096. doi: 10.1016/j.chest.2023.06.029. Epub 2023 Jun 27. PMID 37385337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at different centers in Russia, United States, Canada, Poland and Romania to compare the efficacy, safety and tolerability of two doses of umeclidinium bromide (UMEC) administered once-daily (OD) via a dry powder inhaler, versus placebo.
Pre-assignment Details: Total 421 participants were included in the study.
Groups:
- Placebo QD: Participants received placebo once daily (QD) via the ELLIPTA dry powder inhaler (DPI) for 24 weeks. Participants also received Fluticasone Furoate (FF) 100 micrograms (mcg) once daily as background therapy, in the morning from a separate ELLIPTA DPI for 24 weeks.
- UMEC 31.25 mcg QD: Participants received UMEC 31.25 mcg once daily via the ELLIPTA DPI for 24 weeks. Participants also received FF 100 mcg once daily as background therapy, in the morning from a separate ELLIPTA DPI for 24 weeks.
- UMEC 62.5 mcg QD: Participants received UMEC 62.5 mcg once daily via the ELLIPTA DPI for 24 weeks. Participants also received FF 100 mcg once daily as background therapy, in the morning from a separate ELLIPTA DPI for 24 weeks.
Period: Overall Study
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Started | 143 | 139 | 139
Completed | 137 | 130 | 131
Not Completed | 6 | 9 | 8
Not completed — Withdrawal by Subject | 1 | 5 | 4
Not completed — Investigator Site Closed | 1 | 2 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Study closed/ Terminated | 0 | 0 | 1
Not completed — Met Protocol Withdrawal Criterion | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD | Total
Number analyzed (Participants) | 143 | 139 | 139 | 421
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (13.93) | 48.7 (15.83) | 48.5 (14.21) | 48.8 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 98 | 298
  Male | 37 | 45 | 41 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 10 | 8 | 8 | 26
  Asian; Central/South Asian Heritage | 1 | 1 | 1 | 3
  Asian; East Asian Heritage | 0 | 1 | 0 | 1
  Asian; South East Asian Heritage | 0 | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  White: Arabic/North African Heritage | 0 | 1 | 0 | 1
  White: White/Caucasian/European Heritage | 131 | 126 | 129 | 386
  Black or African American & White | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinic Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 24
Description: FEV1 is measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The highest of 3 technically acceptable measurements were recorded at each Visit. The Baseline value of clinic FEV1 was last acceptable/borderline acceptable (pre-dose) FEV1 value obtained prior to randomized treatment start date. Change from Baseline was calculated as FEV1 value at Week 24 minus FEV1 value at Baseline. Treatment policy estimand was assessed, including all on- and post-treatment data. Intent-to-Treat Population comprised all randomized participants, excluding those who were randomized in error, who did not receive the study drug. Least square (LS) mean and standard error (SE) data is presented. Different participants may have been analyzed at different time points; thus, overall number of participants analyzed reflects everyone in ITT Population without missing covariate information, with Baseline, at least one post-Baseline measurement.
Time Frame: Baseline (Day 1 pre-dose) and Week 24
Population: Intent-to-Treat Population. Participants with available data at Baseline and at least one time point post-Baseline were analyzed. All on- and post-treatment data was included. Different participants may have been analyzed at different time points.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 141 | 136 | 139
Liters | 0.1289 (0.0298) | 0.3046 (0.0304) | 0.3130 (0.0302)
Statistical Analysis 1: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p < 0.001, Mixed-model repeated measures (MMRM); Mean Difference (Net) = 0.1758, 95% CI 2-sided [0.0920 to 0.2595], Standard Error of Mean 0.0426 — UMEC 31.25 mcg versus placebo
Statistical Analysis 2: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p < 0.001, MMRM; Mean Difference (Net) = 0.1841, 95% CI 2-sided [0.1008 to 0.2675], Standard Error of Mean 0.0424 — UMEC 62.5 mcg versus placebo

2. Secondary Outcome: Mean Change From Baseline in Clinic FEV1 at 3 Hours Post Dose at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The highest of 3 technically acceptable measurements were recorded at each Visit. The Baseline value of clinic FEV1 was the last acceptable/borderline acceptable (pre-dose) FEV1 value obtained prior to randomization (either from Visit 2 pre-dose or from Visit 1 pre-bronchodilator). Change from Baseline was calculated as FEV1 value at Week 24 (recorded at 3 hours post dose) minus FEV1 value at Baseline. The analysis only including data collected on-treatment. LS mean change and SE data is presented.
Time Frame: Baseline (Day 1 pre-dose) and Week 24
Population: Intent-to-Treat Population. Only those participants with available on-treatment data at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 133 | 127 | 129
Liters | 0.1768 (0.0318) | 0.3663 (0.0325) | 0.3744 (0.0322)
Statistical Analysis 1: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA); Mean Difference (Net) = 0.1895, 95% CI 2-sided [0.1000 to 0.2789], Standard Error of Mean 0.0455 — UMEC 31.25 mcg vs Placebo
Statistical Analysis 2: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 0.1976, 95% CI 2-sided [0.1086 to 0.2866], Standard Error of Mean 0.0453 — UMEC 62.5 mcg vs Placebo

3. Secondary Outcome: Number of Participants With On-treatment Adverse Events (AE), Non-serious Adverse Events (Non-SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Number of participants with on-treatment AEs and SAEs and serious adverse events (SAE) and common (>=3%)non-SAEs have been reported.
Time Frame: Up to Week 24
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 143 | 139 | 139
Participants
  Any AE | 65 | 73 | 57
  Any SAE | 5 | 4 | 3
  Any non-SAE | 39 | 47 | 33

4. Secondary Outcome: Number of Participants With On-treatment Abnormal Electrocardiograms (ECG) Findings
Description: A single 12-lead ECG and rhythm strip was recorded after measurement of vital signs and spirometry at given time points. All ECG measurements were measured with participants in supine position after >=5 minutes rest. All ECGs were electronically transmitted to an independent and treatment-blinded cardiologist for the measurement. ECG was obtained 15 minutes to 45 minutes after the administration of study treatment. Data for number of participants with abnormal ECG Findings have been reported.
Time Frame: Week 4 and Week 24
Population: Intent-to-Treat Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 143 | 139 | 139
Participants
  Week 4, n=139, 135, 138: number analyzed (Participants) | 139 | 135 | 138
  Week 4, n=139, 135, 138 | 23 | 26 | 35
  Week 24, n=133, 129, 129: number analyzed (Participants) | 133 | 129 | 129
  Week 24, n=133, 129, 129 | 26 | 23 | 39

5. Secondary Outcome: Mean Change From Baseline in On-treatment Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured at every clinic visit, starting at Visit 1, and prior to conducting spirometry. Blood pressure was measured with participant in sitting position after approximately 5 minutes rest. Baseline value was defined as the latest vital signs assessment prior to randomized treatment start, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the value at specified time point. LS mean and SE data is presented. Different participants may have data available at different time points; thus, the overall number of participants analyzed reflects everyone in the ITT Population without missing covariate information and with a Baseline and at least one post-Baseline measurement.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4, 12 and 24
Population: Intent-to-Treat Population. Participants with available data at Baseline and at least one time point post-Baseline were analyzed. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 139 | 137 | 139
Millimeters of mercury
  SBP, Week 4, n=139, 137, 139 | -0.7 (0.70) | 1.1 (0.71) | 0.3 (0.70)
  SBP, Week 12, n=139, 133, 135: number analyzed (Participants) | 139 | 133 | 135
  SBP, Week 12, n=139, 133, 135 | 0.3 (0.78) | -0.2 (0.79) | 0.6 (0.79)
  SBP, Week 24, n=135, 131, 130: number analyzed (Participants) | 135 | 131 | 130
  SBP, Week 24, n=135, 131, 130 | -0.6 (0.77) | 1.1 (0.78) | -0.1 (0.79)
  DBP, Week 4, n=139, 137, 139 | 0.4 (0.55) | 1.2 (0.56) | 0.6 (0.55)
  DBP, Week 12, n=139, 133, 135: number analyzed (Participants) | 139 | 133 | 135
  DBP, Week 12, n=139, 133, 135 | 0.7 (0.57) | 0.2 (0.59) | 1.8 (0.58)
  DBP, Week 24, n=135, 131, 130: number analyzed (Participants) | 135 | 131 | 130
  DBP, Week 24, n=135, 131, 130 | -0.1 (0.57) | 1.6 (0.58) | 1.4 (0.58)
Statistical Analysis 1: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.083, MMRM; Median Difference (Net) = 1.7, 95% CI 2-sided [-0.2 to 3.7], Standard Error of Mean 1.00 — UMEC 31.25 mcg vs Placebo, SBP, Week 4
Statistical Analysis 2: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.636, MMRM; Median Difference (Net) = -0.5, 95% CI 2-sided [-2.7 to 1.7], Standard Error of Mean 1.11 — UMEC 31.25 mcg vs Placebo, SBP, Week 12
Statistical Analysis 3: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.115, MMRM; Mean Difference (Net) = 1.7, 95% CI 2-sided [-0.4 to 3.9], Standard Error of Mean 1.10 — UMEC 31.25 mcg vs Placebo, SBP, Week 24
Statistical Analysis 4: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.336, MMRM; Mean Difference (Net) = 1.0, 95% CI 2-sided [-1.0 to 2.9], Standard Error of Mean 0.99 — UMEC 62.5 mcg vs Placebo, SBP, Week 4
Statistical Analysis 5: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.787, MMRM; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.9 to 2.5], Standard Error of Mean 1.11 — UMEC 62.5 mcg vs Placebo, SBP, Week 12
Statistical Analysis 6: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.625, MMRM; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.6 to 2.7], Standard Error of Mean 1.10 — UMEC 62.5 mcg vs Placebo, SBP, Week 24
Statistical Analysis 7: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.309, MMRM; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.7 to 2.3], Standard Error of Mean 0.79 — UMEC 31.25 mcg vs Placebo, DBP, Week 4
Statistical Analysis 8: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.521, MMRM; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.1 to 1.1], Standard Error of Mean 0.82 — UMEC 31.25 mcg vs Placebo, DBP, Week 12
Statistical Analysis 9: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.047, MMRM; Mean Difference (Net) = 1.6, 95% CI 2-sided [0.0 to 3.2], Standard Error of Mean 0.81 — UMEC 31.25 mcg vs Placebo, DBP, Week 24
Statistical Analysis 10: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.779, MMRM; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.3 to 1.8], Standard Error of Mean 0.78 — UMEC 62.5 mcg versus placebo, DBP, Week 4
Statistical Analysis 11: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.204, MMRM; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.6 to 2.6], Standard Error of Mean 0.82 — UMEC 62.5 mcg versus placebo, DBP, Week 12
Statistical Analysis 12: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.066, MMRM; Mean Difference (Net) = 1.5, 95% CI 2-sided [-0.1 to 3.1], Standard Error of Mean 0.81 — UMEC 62.5 mcg versus placebo, DBP, Week 24

6. Secondary Outcome: Mean Change From Baseline in On-treatment Pulse Rate
Description: Pulse rate was measured at every clinic visit, starting at Visit 1, and prior to conducting spirometry. Pulse rate was measured with participant in sitting position after approximately 5 minutes rest. Baseline value was defined as the latest vital signs assessment prior to randomized treatment start, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the value at specified time point. LS mean and SE data is presented.
Time Frame: Baseline (Day 1 pre-dose), Weeks 4, 12 and 24
Population: Intent-to-Treat Population. Participants with available data at Baseline and at least one time point post-Baseline were analyzed. Participants with data available at the specified time points are represented by (n=X) in the category titles.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
Number analyzed (Participants) | 139 | 137 | 139
Beats per minute
  Week 4, n=139, 137, 139 | -2.3 (0.69) | -1.0 (0.69) | -0.8 (0.69)
  Week 12, n=139, 133, 135: number analyzed (Participants) | 139 | 133 | 135
  Week 12, n=139, 133, 135 | -0.9 (0.59) | -0.3 (0.60) | 0.8 (0.60)
  Week 24, n=135, 131, 130: number analyzed (Participants) | 135 | 131 | 130
  Week 24, n=135, 131, 130 | -1.8 (0.75) | -0.7 (0.76) | 1.5 (0.76)
Statistical Analysis 1: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.195, MMRM; Mean Difference (Net) = 1.3, 95% CI 2-sided [-0.7 to 3.2], Standard Error of Mean 0.97 — UMEC 31.25 mcg vs Placebo, Week 4
Statistical Analysis 2: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.457, MMRM; Mean Difference (Net) = 0.6, 95% CI 2-sided [-1.0 to 2.3], Standard Error of Mean 0.84 — UMEC 31.25 mcg versus Placebo, Week 12
Statistical Analysis 3: Comparison: Placebo QD vs UMEC 31.25 mcg QD; Test type: Superiority; p = 0.300, MMRM; Mean Difference (Net) = 1.1, 95% CI 2-sided [-1.0 to 3.2], Standard Error of Mean 1.07 — UMEC 31.25 mcg versus Placebo, Week 24
Statistical Analysis 4: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.140, MMRM; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.5 to 3.3], Standard Error of Mean 0.97 — UMEC 62.5 mcg versus Placebo, Week 4
Statistical Analysis 5: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.045, MMRM; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.0 to 3.3], Standard Error of Mean 0.84 — UMEC 62.5 mcg versus Placebo, Week 12
Statistical Analysis 6: Comparison: Placebo QD vs UMEC 62.5 mcg QD; Test type: Superiority; p = 0.002, MMRM; Mean Difference (Net) = 3.4, 95% CI 2-sided [1.3 to 5.5], Standard Error of Mean 1.07 — UMEC 62.5 mcg versus Placebo, Week 24

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events and non-serious adverse events were collected up to 25 weeks.
Description: Intent-to-Treat Population was used to collect adverse events.
Arm/Group | Placebo QD | UMEC 31.25 mcg QD | UMEC 62.5 mcg QD
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/139 | 0/139
Serious Adverse Events (participants affected / at risk) | 5/143 | 4/139 | 3/139
Other Adverse Events (participants affected / at risk) | 39/143 | 47/139 | 33/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QD (N=143) | UMEC 31.25 mcg QD (N=139) | UMEC 62.5 mcg QD (N=139)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QD (N=143) | UMEC 31.25 mcg QD (N=139) | UMEC 62.5 mcg QD (N=139)
Nasopharyngitis (Infections and infestations) | 17 (21) | 14 (20) | 13 (15)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (13) | 6 (8)
Respiratory tract infection viral (Infections and infestations) | 5 (5) | 7 (9) | 4 (4)
Headache (Nervous system disorders) | 11 (22) | 9 (14) | 12 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 2 (2)
Toothache (Gastrointestinal disorders) | 4 (5) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03012061/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT03012061/SAP_001.pdf